CLINICAL TRIAL: NCT01143831
Title: Evaluation of Factors II, VII, IX, X, and Proteins C and S, Following High-dose Vitamin K Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephan Moll, MD (Other)
Responsible Party: Sponsor-Investigator, Stephan Moll, MD, Associate Professor, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-1240
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Thrombosis
Keywords: Vitamin K; Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Vitamin K

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All study participants (Experimental): Three blood collections, one at baseline, one two weeks later, and the final blood collection 4 weeks from baseline, after taking Vitamin K orally for 14 days.
  Interventions: Dietary Supplement: Vitamin K, 20mg

INTERVENTIONS:
Dietary Supplement: Vitamin K, 20mg — Subjects will take 20mg vitamin K by mouth in capsule form everyday for 14 continuous days.
  Other Names: Carlson Vitamin K2 Menatetrenone, in 5mg capsules

SUMMARY:
The purpose of this study is to evaluate factor levels of the pro coagulant factors II, VII, IX, X, and the anticoagulant factors protein C and S in healthy volunteers during the intake of elevated levels of vitamin K in order to investigate whether there is any evidence that high dose vitamin K intake increases plasma coagulation factor activity.

DETAILED DESCRIPTION:
1. Recruit 8 male healthy individuals with no prior history of arterial or venous thrombosis (2 each from each of the following age ranges: 20-34, 35-49, 50-64, >65).
2. Visit 1: Measure baseline activity levels of Factor II, Factor VII, Factor IX, Factor X, and levels of D-Dimer, TAT complexes, protein C and S activities. Also measure thrombin generation potential. Collaboration with a research laboratory will be sought to also determine factor VIIa levels.
3. Visit 2: Measure activity of Factor II, Factor VII, Factor IX, Factor X, levels of D-Dimer, TAT complexes, protein C and S activities and thrombin generation potential at the end of the 2 week period.
4. Have each individual consume 20 mg of Vitamin K2 orally per day for two weeks.
5. Visit 3: Measure Factor II, Factor VII, Factor IX, Factor X, D-Dimer, TAT complexes, protein C and S activities and thrombin generation potential at the end of the 2 week period.
6. Total length of study is 4 weeks.
7. Analyze the data sets for changes in levels / activities due to Vitamin K supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male

Exclusion Criteria:

* prior history of arterial or venous thrombosis

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in levels and activities due to vitamin K supplementation | 4 weeks
  Levels and activities to be recorded at three time points: Factor II, Factor VII, Factor IX, Factor X, D-dimer, TAT complexes, Protein C and S, thrombin generation potential

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Moll, MD, Principal Investigator — UNC Chapel Hill Department of Medicine, Division of Hematology
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States